CLINICAL TRIAL: NCT04713137
Title: Effects of Oral Pre-loads on Subsequent Energy Intake, Gastrointestinal Hormones, Glycemic Control, Appetite-related Sensations, and Gastrointestinal Tolerance
Brief Title: Effects of Oral Pre-loads on Subsequent Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PolyFoodIntake
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Energy Intake; Gastrointestinal Hormones; Glycemic Control; Appetite; Satiation
MeSH Terms: interventions — Erythritol; Sucrose; trichlorosucrose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Erythritol (Active Comparator): 20 volunteers receive 50g erythritol dissolved in 300mL tap water as an oral pre-load.
  Interventions: Dietary Supplement: Erythritol
- Sucrose (Active Comparator): 20 volunteers receive 33.5g sucrose dissolved in 300mL tap water as an oral pre-load.
  Interventions: Dietary Supplement: Sucrose
- Sucralose (Active Comparator): 20 volunteers receive 0.0558g sucralose dissolved in 300mL tap water as an oral pre-load.
  Interventions: Dietary Supplement: Sucralose
- Water (Placebo Comparator): 20 volunteers receive 300mL tap water as an oral pre-load.
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Erythritol — 50g erythritol dissolved in 300mL tap water.
  Other Names: E968-Erythritol
  Arms: Erythritol
Dietary Supplement: Sucrose — 33.5g sucrose dissolved in 300mL tap water.
  Other Names: Saccharose
  Arms: Sucrose
Dietary Supplement: Sucralose — 0.0558g sucralose dissolved in 300mL tap water.
  Other Names: E955-Sucralose
  Arms: Sucralose
Dietary Supplement: Water — 300mL tap water.
  Arms: Water

SUMMARY:
The aim of this project is to investigate the effect of erythritol (given as pre-load), compared to sucrose, sucralose, and water on energy intake during a subsequent ad libitum test meal in healthy participants.

Furthermore, the release of GI hormones, glycemic control, appetite-related sensations, GI tolerance, sweetness and liking in response to the pre-loads will be investigated.

DETAILED DESCRIPTION:
The subjects will participate in four study days. The screening will last 60 minutes, the study days about 4.5 hours each. After a simple-carbohydrate standard dinner, the subjects have to do an overnight fast until the next morning. Subjects will receive fixed equisweet doses of sucrose (33.5g), erythritol (50g), sucralose (0.0558g), or water as oral pre-loads in a blinded, randomized (counterbalanced) fashion (t = -15 min). Fifteen minutes after the administration (t = 0 min), a standard solid test meal will be presented and ad libitum calorie intake will be measured. The end of the test meal will be after 20 minutes or as soon as the subject stops eating for more than 5 minutes. Blood samples (to measure: glycemic control and GI hormones) will be collected at t = -16, t = -1, t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 min and appetite-related sensation rating will be collected at t = -16, t = -1, t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 min. GI symptoms and nausea are assessed at t = -16, -1, 30, 60, 120 and 180 min. At t = -10 min subjects are asked to rate the perceived sweetness and liking of the pre-load and at t = 180 min the perceived liking of the test meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal weight subjects with a body-mass index of 19.0-24.9
* Normal eating habits (eating breakfast; no diets; no dietary changes; no vegetarians/vegans, no intolerances/allergies)
* Age 18-55 years
* Stable body weight (+/- 5%) for at least three months
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Shift worker
* Fructose intolerance
* Pre-existing consumption of erythritol and/or sucralose more than once a week
* Substance abuse
* Regular intake of medications, except anticontraceptive
* Chronic or clinically relevant acute infections
* Pregnancy: although no contraindication, pregnancy might influence metabolic state. Women who are pregnant or have the intention to become pregnant during the course of the study are excluded. Female participants of childbearing age have to use safe contraception (oral, injectable, or implantable contraceptives, intrauterine contraceptive devices, or tubectomy). In female participants a urine pregnancy test is carried out upon screening.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Effect of erythritol on energy intake during a subsequent ad libitum test meal | Total energy intake will be measured from t = 0 until t = 20 minutes or as soon as the as the subject stops eating for more than 5 minutes.
  Fifteen minutes after the administration of the pre-loads (t = 0 minutes), a standard solid test meal will be presented and ad libitum calorie intake will be measured.

SECONDARY OUTCOMES:
Effects on GI hormone response - GLP-1 | Blood will be drawn at the following time points: t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Plasma GLP-1 will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA).
Effects on GI hormone response - PYY | Blood will be drawn at the following time points :t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Plasma PYY will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA).
Effects on GI hormone response - CCK | Blood will be drawn at the following time points: t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Plasma cholecystokinin (CCK) levels will be measured with a sensitive radioimmunoassay using a highly specific antiserum.
Effects on GI hormone response - ghrelin | Blood will be drawn at the following time points: t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Plasma ghrelin will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA).
Effects on glycemic control - plasma glucose | Blood will be drawn at the following time points: t = -16, t = -1 (before administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Blood glucose concentrations will be measured by a commercial hexokinase-glucose-6-phosphate-dehydrogenase method (Roche, Basel, Switzerland).
Effects on glycemic control - plasma insulin | Blood will be drawn at the following time points: t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Insulin will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA). The lowest level of insulin that can be detected by this assay is 87 pg/mL when using a 25 µL sample. The intra-assay coefficient of variation for insulin is below 10%, whereas the inter-assay coefficient of variation is below 15%.
Effects on glycemic control - plasma c-peptide | Blood will be drawn at the following time points: t = -16, t = -1 (before administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  C-peptide will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA). The lowest level of c-peptide that can be detected by this assay is 9.5 pg/mL when using a 25 µL sample. The intra-assay coefficient of variation for c-peptide is below 10%, whereas the inter-assay coefficient of variation is below 15%.
Effects on glycemic control - plasma glucagon | Blood will be drawn at the following time points: t = -16, t = -1 (before the administration of the pre-load), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-load).
  Glucagon will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA). The lowest level of glucagon that can be detected by this assay is 13 pg/mL when using a 25 µL sample. The intra-assay coefficient of variation for glucagon is below 10%, whereas the inter-assay coefficient of variation is below 15%.
Effects on appetite-related sensations | Visual analogue scales will be recorded at the following time points: t = -16, t = -1 (before the administration of the pre-loads), t = 15, t = 30, t = 60, t = 90, t = 120, t = 150, t = 180 minutes (after the administration of the pre-loads).
  Appetite perceptions (feelings of: a) hunger, b) satiety) are assessed by visual analogue scale (VAS). Visual analogue scales consist of a horizontal, unstructured, 10-cm line representing the minimum (0.0 points) to the maximum rating (10.0 points). Subjects assign a vertical mark across the line to indicate the magnitude of their subjective sensation at the present time point. The measurement is quantified by the distance from the left end of the line (minimum rating) to the subject's vertical mark.
Effects on GI tolerance | GI tolerance will be recorded at t = -16, -1 (before the administration of the pre-load), 30, 60, 120 and 180 minutes (after the administration of the pre-load).
  GI symptoms will be assessed by use of a checklist including the following questions: abdominal pain, nausea, vomiting, diarrhoea, borborygmi, abdominal distension, eructation and increased flatus.
Sweetness of pre-load | Sweetness of the pre-load will be recorded at t = -10 minutes.
  Sweetness is assessed by gLMS. General Labeled Magnitude Scales consist of an unequal, vertical line, which is marked with quasi-logarithmic verbal anchors describing different intensities (e.g. "strongest imaginable", "barely detectable"). Participants are instructed to place a mark on the line where their perceived intensity of sensation lies.
Liking ot the pre-load | Liking of the pre-load will be recorded at t = -10 minutes.
  Liking is assessed by gLMS. General Labeled Magnitude Scales consist of an unequal, vertical line, which is marked with quasi-logarithmic verbal anchors describing different intensities (e.g. "strongest imaginable", "barely detectable"). Participants are instructed to place a mark on the line where their perceived intensity of sensation lies.
Liking of the test meal | Liking of the test meal will be recorded at t = 180 minutes.
  Liking is assessed by gLMS. General Labeled Magnitude Scales consist of an unequal, vertical line, which is marked with quasi-logarithmic verbal anchors describing different intensities (e.g. "strongest imaginable", "barely detectable"). Participants are instructed to place a mark on the line where their perceived intensity of sensation lies.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Christin Meyer-Gerspach, PD, PhD, Principal Investigator — St. Clara Research Ltd.
Locations (1):
- St. Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No